CLINICAL TRIAL: NCT04069910
Title: Neoadjuvant Stereotactic Radiation Therapy for Resectable Brain Metastases
Brief Title: Stereotactic Radiation Therapy Before Surgery for the Treatment of Resectable Brain Metastases
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enrollment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-000082; NCI-2019-05337 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2020-09

CONDITIONS: Malignant Neoplasm, Brain; Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm A (SRS/SRT, surgery) (Experimental): Patients undergo 1, 5, or 10 fraction of SRS/SRT radiation. Surgery is performed within 72 hours of radiation therapy.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery; Procedure: Therapeutic Conventional Surgery
- Arm B (surgery, SRS/SRT) (Active Comparator): Within 2-5 weeks after standard of care surgery, patients undergo 1, 5, or 10 fraction of SRS/SRT.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Radiosurgery — Undergo SRS/SRT
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; stereotactic radiation therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgery

SUMMARY:
This trial studies how well stereotactic radiation therapy before surgery works in treating patients with cancer that has spread to the brain (brain metastases) and can be removed by surgery (resectable). Stereotactic radiation therapy is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor, and may cause less damage to normal tissue. Giving stereotactic radiation therapy before surgery may make the return of brain metastases less likely and help patients live longer compared to surgery followed by radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rate of leptomeningeal failure after neoadjuvant radiation therapy (NaRT) versus (vs) postoperative stereotactic radiosurgery (SRS)/stereotactic radiation therapy (SRT).

SECONDARY OBJECTIVES:

I. Local control of brain metastases. II. Rate of salvage treatment including surgery, SRS, SRT, or whole brain radiation therapy (WBRT).

III. Dose and volume of radiation to adjacent normal brain parenchyma. IV. Rate of symptomatic radiation necrosis/steroid dependency. V. Rate of distant brain failure. VI. To compare overall survival (OS) between the 2 groups. VII. To determine the number of patients who die due to neurologic causes. VIII. To assess quality of life as assessed using Functional Assessment of Cancer Therapy?Brain (FACT?BR).

IX. To evaluate and compare the molecular makeup of tumor tissue in pre vs post radiation settings and determine differences in molecular and germline markers.

X. To evaluate biomarkers and germline markers predicting response.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo 1, 5, or 10 fraction of SRS/SRT radiation. Surgery is performed within 72 hours of radiation therapy.

ARM B: Within 2-5 weeks after standard of care surgery, patients undergo 1, 5, or 10 fraction of SRS/SRT.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Prior histologic diagnosis of cancer other than small cell lung cancer, lymphoma, and germ cell histologies
* 1?4 cerebral metastases per magnetic resonance imaging (MRI) with at least 1 being dominant and eligible for resection
* No prior radiation treatment for the index brain metastases
* Systemic disease staged within previous 8 weeks and not rapidly progressing, with concern of life expectancy > 3 months
* The patients will have been evaluated by the multidisciplinary team, and surgery must be deemed necessary as a result of indications including but not limited to mass effect or symptomatic lesion. Surgery must be deemed non?emergent or non?urgent clinically by the neurosurgeon
* Karnofsky performance status (KPS) >= 70
* No active infections requiring systemic antibiotics
* If a woman is of childbearing potential, a negative serum pregnancy test must be documented. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) for duration of study participation and for up to 4 weeks following the study treatment
* Ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* Patient deemed medically unfit to undergo surgical resection of brain metastasis
* Prior whole brain radiotherapy
* Patient with contraindication for imaging with MRI
* Surgery is considered emergent or urgent by the neurosurgeon due to symptoms or concerning mass effect noted on imaging
* Patients who are participating in a concurrent treatment protocol
* At the time of planning, unable to meet dose tolerance of the optic nerve/chiasm
* Tumor located in the brainstem
* Imaging or cytologic evidence of leptomeningeal disease
* Concurrent uncontrolled illness including, but not limited to, any of the following: Symptomatic congestive heart failure, unstable angina pectoris, psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of leptomeningeal failure | Up to 2 years
  A two-sided Z test with pooled variance will be used at significance level =0.1 to test if there is a difference in leptomeningeal failure rate between the two treatment groups.

SECONDARY OUTCOMES:
Time to progression | Up to 2 years
  Local control of brain metastases is defined as tumor has not progressed or recurred with no radiographic or symptomatic progression. Using the Response Assessment in Neuro-Oncology (RANO) criteria for brain metastases, progressive disease will be defined as > 20% increase in the sum of the longest diameters of the target lesions; unequivocal progression of enhancing non?target lesions; new lesions; or substantial clinical decline. Will be compared using t test for continuous outcomes, log rank test for time?to?event outcomes and Z test for binary outcomes.
Rate of salvage treatment including surgery, SRS, SRT, or WBRT | Up to 2 years
  Will be compared using t test for continuous outcomes, log rank test for time?to?event outcomes and Z test for binary outcomes.
Dose (Gy) and volume (cc) of radiation to adjacent normal brain parenchyma | Up to 2 years
  Will be compared using t test for continuous outcomes, log rank test for time-to-event outcomes and Z test for binary outcomes.
Rate of symptomatic radiation necrosis/steroid dependency | Up to 2 years
  Will be compared using t test for continuous outcomes, log rank test for time?to?event outcomes and Z test for binary outcomes.
Rate of distant brain failure | Up to 2 years
  Will be compared using t test for continuous outcomes, log rank test for time?to?event outcomes and Z test for binary outcomes.
Overall survival (OS) | Up to 2 years
  Will be compared using t test for continuous outcomes, log rank test for time?to?event outcomes and Z test for binary outcomes.
Death due to neurological causes | Up to 2 years
  Will be compared using t test for continuous outcomes, log rank test for time?to?event outcomes and Z test for binary outcomes.
Quality of life assessment: FACTBR | Up to 2 years
  Assessed using Functional Assessment of Cancer Therapy-Brain (FACTBR). Will be compared using t test for continuous outcomes, log rank test for time?to?event outcomes and Z test for binary outcomes. The scale is 0 - 4, 0 = "not at all", 4 = "very much". Overall higher ratings mean higher quality of life.
Genetic expression profiles in pre vs post radiation tumor tissue | Up to 2 years
  Will be compared using t test for continuous outcomes, log rank test for time?to?event outcomes and Z test for binary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Tania B Kaprealian, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States